CLINICAL TRIAL: NCT03254212
Title: Evaluation of Nocturnal Oxygen Needs in the Treatment of Central Sleep Apnea in Patients With Chronic Heart Failure.
Brief Title: Nocturnal Oxygen Needs and Central Sleep Apnea in Patients With Chronic Heart Failure.
Acronym: HO2F
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Oxynov (Unknown); Philips Respironics (Industry)
Responsible Party: Principal Investigator, Frédéric Sériès, Director IUCPQ Sleep laboratory, Laval University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OXY-GRA-17027-LOFTHF-SH
Record Dates: First submitted 2017-07-25; First posted 2017-08-18 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Chronic Heart Failure; Central Sleep Apnea
Keywords: Heart failure; Central sleep apnea; oxygen therapy
MeSH Terms: conditions — Sleep Apnea, Central; Heart Failure

STUDY DESIGN:
Intervention Model Description: Fixed nightime oxygen therapy throughout the study duration with oxygen flow determined according to the results of the home oxygen titration procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxygen therapy (Experimental): Fixed nightime oxygen therapy throughout the protocol duration
  Interventions: Device: Titration of nocturnal oxygen needs to prevent desaturations

INTERVENTIONS:
Device: Titration of nocturnal oxygen needs to prevent desaturations — Oximetry recordings will be performed using a Pulse Oximeter. Two O2 titration sessions will be conducted at home in random order one week apart. One will consist of a stepwise night-to-night increase in O2 flow for up to 4 nights with supplemental O2, each at flow rates of 1L/min, 2L/min, 3L/min and 4L/min, respectively. During the other titration session, an automatic O2 delivery system will be used for 4 consecutive nights with O2 flow allowed to vary from 0 to 4 L/min with a 95 ± 2% SpO2 target. At the end of the titration periods, oxygen concentrators will be set at the lowest flow rate (1L/min to 4L/min) that maintained oxyhemoglobin saturation to > 90% (Tsat90%) for ≥ 98% of the estimated sleep period and reduced the oxygen desaturation index 3% (ODI3) to < 5/hour according to conventional O2 titration. If these targets are not reached, the lowest flow rate will be selected that minimizes the ODI3. These procedures will be repeated at week 5 and 11.

SUMMARY:
The aims of this study are to 1) determine the optimal levels of O2 flow which prevent nocturnal O2 desaturation while minimizing periods of hyperoxia during the course of nocturnal oxygen therapy (NOXT) in heart failure patients with reduced ejection fraction (HFrEF) patients with CSA/CSR; 2) document whether within-patient EO2F values change over time during NOXT, and identify factors which predict changes in EO2F; and 3) examine how well a conventional stepwise titration procedure compares to a breath by breath titration using an automated O2 titration system in terms of targeted flow rate and night time oxygenation (oxygen desaturation index, time spent at specific SpO2 targets).

DETAILED DESCRIPTION:
Sleep-related breathing disorders (obstructive and central) are highly prevalent in Heart failure (HF) patients and are associated with an increase in morbidity and mortality. Nocturnal oxygen therapy (NOT) reduces the frequency of central breathing events by 75 % and prevents nocturnal desaturation in patients with HF. Considering that the amount of nocturnal desaturation is a better predictor of mortality than the apnea+hypopnea index (AHI) in this population, one should expect NOT to have a positive impact on survival in these patients. In the four randomized clinical trials where the effects of O2 on left ventricular function was assessed, 2 reported a significant increase in LVEF after 3 months of NOT. NOT was also found to positively impact on other important predictive factors of mortality such as sympathetic activity and VO2 max. These mitigated results could be accounted by the fact that a fixed O2 flow was empirically used (2 to 4 L/min) in the majority of studies. This may impede the beneficial effects of NOT for two reasons. First, in patients with HF, oxygen is associated with a dose-related detrimental hemodynamic effects (i.e. increase in vascular resistance and reduction in cardiac output and stroke volume). Therefore, the lowest O2 flow that prevents nocturnal desaturation should be used to minimize the detrimental effects of hyperoxia. On the other hand, there are evidences that the frequency and/or severity of sleep-disordered breathing may change overtime in CHF patients leading to insufficient correction of nocturnal desaturation during the course of NOT. Therefore, NOT should be preceded by an oxygen titration procedure to determine the lowest O2 flow that prevents nocturnal desaturation. This can be done with a stepwise night-to-night increase in O2 flow until correction of nocturnal desaturation. However, another approach would be to prevent event-by-event desaturations and to prevent hyperoxia during periods of normal sleep and wakefulness. On the other hand, the stability in O2 needs overtime in these patients is unkown. The aims of this study are 1) to document if the level of O2 flow preventing nocturnal desaturation changes during the course of NOT in CHF patients with CSA/CSR and 2) to examine the ability of automated O2 titration (FreeO2, Oxynov, Quebec, Canada) to determine O2 needs in HF patients with CSA/CSR when compared to the gold standard titration procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients with heart failure and reduced ejection fraction (LVEF < 45%) due to ischemic or hypertensive heart disease
* moderate to severe central sleep apnea/cheyne stokes respiration.
* treatment should be stable for the last 30 days preceding entry into the study.

Exclusion Criteria:

* O2 /CPAP therapy,
* active smoking,
* primary valvular heart disease,
* nasal obstruction,
* BMI ≥ 32 Kg/m2,
* cardiac surgery/transient ischemic attack/stroke/resynchronization therapy within 3 months,
* nocturnal hypoventilation,
* receiving opiates or methadone medication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in optimal levels of O2 flow ( EO2F) which prevent nocturnal O2 desaturation | Three months ( titration completed 3 times during the study period)
  changes in the lowest flow rate (1L/min to 4L/min) that maintained oxyhemoglobin saturation to > 90% (Tsat90%) for ≥ 98% of the estimated sleep period and reduced the oxygen desaturation index (ODI3P) to < 5/hour
Accuracy of automated oxygen titration | Three months (new titration sessions completed 3 times during the study period)
  examine how well a conventional stepwise titration procedure compares to a breath by breath titration using an automated O2 titration system in terms of targeted flow rate and night time oxygenation (oxygen desaturation index, time spent at specific SpO2 targets)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Frédéric Sériès, Québec, Qiebec
  - John Kimoff, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No